CLINICAL TRIAL: NCT02777632
Title: Resistant Bacterial Infections in the Early Post LDLT Period
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Mahmoud Aly Massoud, Lecturer of Tropical medicine, Ain Shams University
Other Study IDs: 2652010
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Transplantation Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- HCV patients following living donor liver transplantation: single infection episode group
  Interventions: Procedure: Living donor liver transplantation
- patients following living donor liver transplantation: recurrent Infections episode group
  Interventions: Procedure: Living donor liver transplantation

INTERVENTIONS:
Procedure: Living donor liver transplantation

SUMMARY:
The purpose of this work was to study the incidence, types, risk factors and causative organisms of bacterial infections in HCV Egyptian patients following Liver Transplantation. Moreover, to identify the emerging resistant strains and their proper antimicrobial therapy

DETAILED DESCRIPTION:
This prospective descriptive study has been done at Tropical Medicine department in the period between January 2014 to November 2015.

After the approval of the scientific and ethical committee of Ain Shams University Hospital, Patients with HCV positive end stage liver disease (ESLD) eligible for liver transplantation Ain Shams Center for Organ Transplant (ASCOT); Ain Shams University, (fulfilling the inclusion criteria) were included in the current study. Forty five patients were recruited and each one was followed-up during a period of 3 months following transplantation.

Included patients were divided into 2 groups:

Group 1 included patients who had a postoperative single episode of infection. Group 2 included those patients who had more than 1 episode of postoperative bacterial infection whom were further evaluated for the presence of emerging strains and/or antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian nationality.
* Accepting participation in the current study and signing a written consent form
* Age between 18-60 Years, including males and females.

Exclusion Criteria:

* Patients who refused to be enrolled in the study.
* Patients with other etiologies for end-stage liver disease (HBV, PBC…)
* Patients with preoperative infections, infections within 48 h after transplantation or early post-operative death

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HCV patients who underwent living donor liver transplantation at Ain Shams Center for Organ Transplantation.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Determine the types of early bacterial infections following LDLT, recurrent and resistant infections all were confirmed by cultures. | Within the first 90 days after the operation
  Bile, abdominal drains, blood stream infection, urinary tract infection or chest infection.
Assessment of risk factors for occurrence of recurrent bacterial infections | The first 3 months following LDLT
  Independent risk factors for infections

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine M Massoud, MD, Principal Investigator — Faculty of Medicine, Ain Shams University